CLINICAL TRIAL: NCT01772420
Title: Phase II Study of Lenalidomide and Eltrombopag in Patients With Symptomatic Anemia in Low or Intermediate I Myelodysplastic Syndrome (MDS)
Brief Title: Phase II Study of Lenalidomide and Eltrombopag in Patients With Symptomatic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-407; NCI-2013-01219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA013330 (NIH); 115479 (Other: GlaxoSmithKline Tracking Number); RV--MDS-PI-0645 (Other: Celgene Tracking Number)
Record Dates: First submitted 2013-01-15; First posted 2013-01-21 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Adult Myelodysplastic Syndrome; Anemia; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Anemia; Leukemia, Myelomonocytic, Chronic | interventions — eltrombopag; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (lenalidomide, eltrombopag olamine) (Experimental): Patients with baseline platelet counts >= 50,000 receive lenalidomide PO daily or QOD on days 1-21. If platelet counts fall below 50,000, patients discontinue lenalidomide and receive eltrombopag olamine PO daily or QOD until platelet count is maintained above 50,000 for 2 weeks. Patients then resume lenalidomide PO daily or QOD. If platelets fall below 50,000 again, patients receive eltrombopag olamine as before. When platelet counts are maintained above 50,000 for 2 weeks, patients resume lenalidomide concurrently with eltrombopag for all subsequent courses.
  Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eltrombopag Olamine; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm B (eltrombopag olamine, lenalidomide) (Experimental): Patients with baseline platelet counts < 50,000 receive eltrombopag olamine PO daily or QOD on days 1-28 until platelet count is maintained above 50,000 for 2 weeks. Patients then receive treatment as in Arm A.
  Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eltrombopag Olamine; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Drug: Eltrombopag Olamine — Given PO
  Other Names: Promacta; SB-497115-GR
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial studies how well lenalidomide (LEN) and eltrombopag olamine (ELT) work in treating patients with symptomatic anemia in low or intermediate myelodysplastic syndrome (MDS). Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. Eltrombopag olamine may increase the number of white blood cells and platelets found in bone marrow or peripheral blood. Giving lenalidomide and eltrombopag olamine may be an effective treatment for myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES (not Outcome Measures):

I. To evaluate the rate of hematologic improvement of the eltrombopag (eltrombopag olamine)/lenalidomide combination (as per Modified International Working Group [IWG] criteria).

II. To evaluate the safety and tolerability of the combination.

SECONDARY OBJECTIVES (not Outcome Measures):

I. To compare the time to hematologic improvement. II. To evaluate the duration of hematologic improvement III. To evaluate the effect of combination treatment on platelet counts, platelet transfusions and bleeding events.

IV. To evaluate the frequency of bone marrow response (complete response [CR] + partial response [PR]) and cytogenetic response.

V. To evaluate the relationship between mutations in bone marrow stem cells and response.

VI. To evaluate the relationship between various stem and progenitor alterations and response.

OUTLINE: Patients are initially assigned to 1 of 2 treatment arms.

ARM A: Patients with platelet counts >= 50,000 receive lenalidomide orally (PO) daily or every other day (QOD) on days 1-21. If platelet counts fall below 50,000, patients discontinue lenalidomide and receive eltrombopag olamine PO daily or QOD until platelet count is maintained above 50,000 for 2 weeks. Patients then resume lenalidomide PO daily or QOD. If platelets fall below 50,000 again, patients receive eltrombopag olamine as before. When platelet counts are maintained above 50,000 for 2 weeks, patients resume lenalidomide concurrently with eltrombopag for all subsequent courses.

ARM B: Patients with platelet counts < 50,000 receive eltrombopag olamine PO daily or QOD on days 1-28 until platelet counts is maintained above 50,000 for 2 weeks. Patients then receive treatment as in Arm A.

In both arms, treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 5 years.

Eligible patients with a diagnosis of MDS or non-proliferative chronic myelomonocytic leukemia (CMML) (WBC ≤ 12,000/mL) of at least 3-month duration according to WHO criteria and International Prognostic Scoring System categories of low or intermediate-1-risk disease. Patients either had symptomatic anemia untransfused with hemoglobin ≤ 10 g/dL in the 8 weeks before starting the study or had RBC transfusion dependence (i.e., ≥ 2 units/mo) confirmed 8 weeks before starting the study and/or PLTs <50,000 k/uL with hemoglobin >10.0 g/dL. Patients must not have received prior therapy with LEN (for > 2 months) nor ELT

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a documented diagnosis of myelodysplastic syndrome (MDS) of at least three months duration (MDS duration >= 3 months) according to World Health Organization (WHO) criteria or non-proliferative chronic myelomonocytic leukemia (CMML) (white blood cells [WBC] =< 12,000/L)
* Patients must have International Prognostic Scoring System (IPSS) categories of low- or intermediate-1-risk disease
* Patients must have symptomatic anemia untransfused with hemoglobin =< 9.5 g/dL within 8 weeks of registration or with red blood cell (RBC) transfusion-dependence (i.e., >= 2 units/month) confirmed for a minimum of 8 weeks before randomization
* Patients must have IPSS score determined by cytogenetic analysis prior to randomization; patients with cytogenetic failure and =< 10% marrow blasts will be eligible
* Patients must be off all disease modifying therapy for MDS for 28 days prior to initiation of study treatment; patients may receive hydrocortisone prophylactically to prevent transfusion reactions
* Patients must not have documented iron deficiency; all patients must have documented marrow iron stores; if marrow iron stain is not available, the transferrin saturation must be >= 20% or a serum ferritin >= 100 ng/100 mL or soluble transferring receptor < 5 mg/L.
* Women must not be pregnant or breastfeeding; females of childbearing potential should have 2 negative pregnancy tests (sensitivity of at least 50 mIU/mL); the first test should be performed within 10-14 days, and the second test within 24 hours prior to prescribing lenalidomide
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program; able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin)
* Women of childbearing potential and sexually active males must agree to use 2 methods of an accepted and effective method of contraception and counseled on the potential teratogenic effects of lenalidomide; effective contraception must be used by patients for at least 4 weeks before beginning lenalidomide therapy, during lenalidomide therapy, during dose interruptions and for 4 weeks following discontinuation of lenalidomide therapy; reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or because the patient has been postmenopausal naturally for at least 24 consecutive months; two reliable forms of contraception must be used simultaneously unless continuous abstinence from heterosexual sexual contact is the chosen method; females of childbearing potential should be referred to a qualified provider of contraceptive methods, if needed; sexually mature females who have not undergone a hysterectomy or who have not been postmenopausal naturally for at least 24 consecutive months (i.e., who have had menses at some time in the preceding 24 consecutive months) are considered to be females of childbearing potential; it is not known whether CC-5013 (lenalidomide) is present in the semen of patients receiving the drug; therefore, males receiving CC-5013 (lenalidomide) must always use a latex condom during any sexual contact with females of childbearing potential even if they have undergone a successful vasectomy
* Patients must not have received prior therapy with lenalidomide (for more than 2 months) nor eltrombopag
* Patients must not have uncontrolled hypertension
* Patients must have absolute neutrophil count (ANC) >= 500 cells/L (0.5 x 10^9/L)
* Eastern Cooperative Oncology Group (ECOG) performance 0-3
* Subject is able to understand and comply with protocol requirements and instructions
* Patient has signed and dated informed consent
* Prothrombin time (PT/international normalized ratio [INR]) and activated partial thromboplastin time (aPTT) must be within 80 to 120% of the normal range at baseline

Exclusion Criteria:

* Pre-existing cardiovascular disease (including congestive heart failure, New York Heart Association [NYHA] grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a corrected QT interval (QTc) > 450 msec
* Patients determined to be at increased risk of arterial or venous thrombosis by the investigator
* Bone marrow fibrosis that leads to a dry tap
* Female subjects who are nursing or pregnant (positive serum or urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test) at screening or pre-dose on day 1
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
* Patients with documented liver cirrhosis
* Patients with splenomegaly with a spleen size > 16 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-10; Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit K Verma, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Albert Einstein College of Medicine, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From October 2012 through January 2020, 52 patients were enrolled in this multicenter study.
Groups:
- Arm A (Platelets > 50,000 k/uL) LEN Initiation: Patients with baseline platelet counts >50,000 k/uL received lenalidomide (LEN) PO daily or QOD on days 1-21. If platelet counts fell below 50,000 k/uL during treatment, patients discontinued LEN and received eltrombopag olamine (ELT) PO daily or QOD until platelet counts > 50,000 k/uL were achieved, and then maintained for 2 weeks thereafter. If a platelet count >50,000 k/uL was maintained, patients discontinued ELT and resumed only LEN as a single agent (PO daily or QOD). If platelets fell below 50,000 k/uL a second time, LEN was stopped and ELT was re-initiated at the dose last given to the patient. Once platelet counts were >50,000 k/uL and maintained for 2 weeks, patients resumed LEN concurrently with ELT for all subsequent courses.
  Treatment repeated every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Eltrombopag Olamine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
- Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination: Patients with baseline platelet counts <50,000 k/uL received eltrombopag olamine (ELT) PO daily or QOD on days 1-28 until a platelet count >50,000 k/uL was achieved. Once a platelet count>50,000 k/uL was achieved the ELT dose was maintained for two weeks. After two weeks ELT was discontinued and LEN was started as in Arm A (i.e., eltrombopag olamine discontinued and lenalidomide started). Patients in Arm B were permitted to stay on ELT alone if a hematologic response on ELT was achieved as defined by the 2006 International Working Group (IWG) consensus criteria, or if baseline hemoglobin was >10.0 g/dL and didn't decrease while on study drug.
  Treatment repeated every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Eltrombopag Olamine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
- Arm C (Platelets < 50,000 k/uL) ELT Monotherapy: Patients in Arm B were permitted to stay on ELT alone if a hematologic response on ELT was achieved as defined by the 2006 International Working Group (IWG) consensus criteria, or if baseline hemoglobin was >10.0 g/dL and didn't decrease while on study drug.
  Treatment repeated every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Eltrombopag Olamine: Given PO Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Started | 16 | 15 | 21
Completed | 16 | 15 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy | Total
Number analyzed (Participants) | 16 | 15 | 21 | 52
Age, Continuous [Mean (Full Range); unit: years] | 74 [59 to 86] | 73 [56 to 85] | 68 [34 to 93] | 71 [34 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 4 | 15
  Male | 9 | 11 | 17 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 11 | 10 | 8 | 29
  Non-Hispanic Black | 1 | 1 | 7 | 9
  Hispanic | 4 | 4 | 3 | 11
  Asian | 0 | 0 | 2 | 2
  Unknown (Not Documented) | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 21 | 52
Baseline Hemoglobin [Mean (Full Range); unit: g/dL] | 8.2 [6.2 to 9.5] | 8.1 [6.4 to 10.8] | 8.6 [6.1 to 11.7] | 8.4 [6.1 to 11.7]
Baseline Platelet [Mean (Full Range); unit: platelets x10^9/L] | 257 [88 to 457] | 134 [16 to 280] | 19 [1 to 97] | 126 [1 to 457]
Blast Count [Mean (Full Range); unit: percentage of blasts in bone marrow cell] | 1.96 [0 to 5] | 1.87 [0 to 6] | 1.8 [0 to 8] | 1.87 [0 to 8]
Myelodysplastic Syndrome (MDS) [Count of Participants; unit: Participants] | 16 | 14 | 19 | 49
Chronic Myelomonocytic Leukemia (CMML) [Count of Participants; unit: Participants] | 0 | 1 | 2 | 3
Revised International Prognostic Scoring System (IPSS-R) for Myelodysplastic Syndrome (MDS) [Count of Participants; unit: Participants]
  Very Low Risk | 1 | 0 | 0 | 1
  Low Risk | 8 | 10 | 6 | 24
  Intermediate Risk | 7 | 5 | 15 | 27
Number of Prior Treatments [Mean (Full Range); unit: Prior Treatments] | 0.63 [0 to 3] | 0.53 [0 to 2] | 0.48 [0 to 3] | 0.54 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Demonstrating Overall Hematologic Improvement (HI)
Description: The number of patients demonstrating overall Hematologic Improvement (HI) was assessed based on the MDS 2006 IWG criteria. The IWG criteria for HI define specific responses of cytopenia in the 3 hematopoietic lineages: erythroid (HI-E), platelet (HI-P), and neutrophil (HI-N) as demonstrated in corresponding outcome measures. Responses must have sustained for at minimum of 8 weeks for the participant to be included in the tally.
Time Frame: Periodic evaluation (weekly up to a month, followed by 4x28 day cycles = 16weeks) with additional cycles and titrations depending upon treatment response; up to 2 years
Population: Intention to treat population study design.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Number analyzed (Participants) | 16 | 15 | 21
Participants | 6 | 5 | 7

2. Secondary Outcome: Number of Patients With Hematologic Improvement in Platelet Counts (HI-P)
Description: The Number of Patients with Hematologic Improvement in Platelet Counts (HI-P) was assessed based on the MDS 2006 IWG criteria. Patients demonstrating an absolute increase of ≥ 30 × 10^9/L (for those patients starting with > 20 × 10^9/L platelets) or an increase from < 20 × 10^9/L to > 20 × 10^9/L along with an increase of at least 100%, were deemed to have demonstrated HI-P improvement.
Time Frame: as for outcome 1
Population: Intention to treat population study design.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Number analyzed (Participants) | 16 | 15 | 21
Participants | 0 | 3 | 6

3. Secondary Outcome: Number of Patients With Hematologic Improvement in Erythrocyte Counts (HI-E)
Description: The Number of Patients with Hematologic Improvement in Erythrocyte Counts (HI-E) was assessed based on the MDS 2006 IWG criteria. Patients demonstrating an Hgb increase by ≥ 1.5 g/dL were deemed to have improvement in HI-E. Only transfusions given for a Hgb of ≤ 9.0 g/dL pretreatment were counted in the RBC transfusion response.
Time Frame: as for outcome 1
Population: Intention to treat population study design.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Number analyzed (Participants) | 16 | 15 | 21
Participants | 6 | 3 | 4

4. Secondary Outcome: Number of Patients With Hematologic Improvement in Neutrophil Counts (HI-N)
Description: The Number of Patients with Hematologic Improvement in Neutrophil Counts (HI-N) was assessed based on the MDS 2006 IWG criteria. Patients demonstrating an increase of at least 100% and an absolute increase > 0.5 × 10^9/L were determined to have shown an improvement in HI-N.
Time Frame: as for outcome 1
Population: Intention to treat population study design.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Number analyzed (Participants) | 16 | 15 | 21
Participants | 0 | 1 | 2

5. Secondary Outcome: Time to Attain Hematologic Improvement (HI)
Description: Time to hematologic improvement as determined by median time required to achieve HI response.
Time Frame: as for outcome 1
Population: Intention to treat population study design.
Measure: Median (Full Range); unit: number of weeks
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Number analyzed (Participants) | 16 | 15 | 21
number of weeks | 12 [2.4 to 16] | 8 [2 to 20] | 8 [6 to 12.4]

6. Secondary Outcome: Duration of Hematologic Improvement (HI)
Description: Duration to hematologic improvement as determined by median duration of HI response.
Time Frame: Time to progression/relapse following hematologic improvement, at completion of final cycle and treatment discontinuation; up to 6 years
Population: Intention to treat population study design.
Measure: Median (Full Range); unit: number of weeks
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Number analyzed (Participants) | 16 | 15 | 21
number of weeks | 41 [25 to 141] | 88 [8.3 to 107] | 40 [8 to 295]

7. Secondary Outcome: Number of Patients With Clinically Significant Bleeding Events
Description: Number of Patients With Clinically Significant Bleeding Events
Time Frame: Treatment initiation through study completion, up to 2 years
Population: Intention to treat population study design.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination: Patients with baseline platelet counts <50,000 k/uL received eltrombopag olamine (ELT) PO daily or QOD on days 1-28 until a platelet count >50,000 k/uL was achieved. Once a platelet count >50,000 k/uL was achieved the ELT dose was maintained for two weeks. After two weeks ELT was discontinued and LEN was started as in Arm A (i.e., eltrombopag olamine discontinued and lenalidomide started). Patients in Arm B were permitted to stay on ELT alone if a hematologic response on ELT was achieved as defined by the 2006 International Working Group (IWG) consensus criteria, or if baseline hemoglobin was >10.0 g/dL and didn't decrease while on study drug.
  Treatment repeated every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Eltrombopag Olamine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
Number analyzed (Participants) | 16 | 15 | 21
Participants | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, up to 2 years
Description: Adverse events categorized based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Groups:
- Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination: Patients with baseline platelet counts <50,000 k/uL received eltrombopag olamine (ELT) PO daily or QOD on days 1-28 until a platelet count >50,000 k/uL was achieved. Once a platelet count>50,000 k/uL was achieved the ELT dose was maintained for two weeks. After two weeks ELT was discontinued and LEN was started as in Arm A (i.e., eltrombopag olamine discontinued and lenalidomide started). Patients in Arm B were permitted to stay on ELT alone if a hematologic response on ELT was achieved as defined by the 2006 International Working Group (IWG) consensus criteria, or if baseline hemoglobin was >10.0 g/dL and didn't decrease while on study drug.
  Treatment repeated every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Eltrombopag Olamine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO Treatment repeated every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Eltrombopag Olamine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
Arm/Group | Arm A (Platelets > 50,000 k/uL) LEN Initiation | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy
All-Cause Mortality (participants affected / at risk) | 1/16 | 2/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 8/16 | 5/15 | 0/21
Other Adverse Events (participants affected / at risk) | 15/16 | 9/15 | 4/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Platelets > 50,000 k/uL) LEN Initiation (N=16) | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination (N=15) | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy (N=21)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (severe) (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) — Severe thrombocytopenia
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Pneumonia
Gall Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Platelets > 50,000 k/uL) LEN Initiation (N=16) | Arm B (Platelets < 50,000 k/uL) ELT Initiation With Potential LEN Combination (N=15) | Arm C (Platelets < 50,000 k/uL) ELT Monotherapy (N=21)
Blood Bilirubin Increased (Investigations) | 0 (0) | 2 (2) | 1 (1) — Hyperbilirubinemia from development of bone marrow fibrosis
Acute Cholecystitis (Investigations) | 2 (2) | 0 (0) | 1 (1) — AST/ALT elevation, reversible increase in peripheral blasts
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Right Arm Hematoma
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT01772420/Prot_SAP_000.pdf